CLINICAL TRIAL: NCT05198726
Title: Speed of Processing (SoP) Training Plus α-tACS in People With Mild Cognitive Impairment: a Double Blind, Parallel, Placebo Controlled Trial Study Protocol
Brief Title: Speed of Processing (SoP) Training Plus α-tACS
Acronym: aMCIUp
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was halted due to the COVID19, and then due to the lack of funding to continue the study
Sponsor: Portucalense University (Other)
Collaborators: Aveiro University (Other); University of Coimbra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UPT01
Record Dates: First submitted 2021-12-20; First posted 2022-01-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cognitive Dysfunction; Mild Cognitive Impairment; tACS; Cognitive Training
Keywords: MCI; tACS; Cognitive training
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: double-blinded, parallel randomized trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Sham tACS and cognitive training
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active tACS plus active SoP (Active Comparator): Active alpha range tACS plus Speed of Processing Training
  Interventions: Device: alpha tACS; Behavioral: Speed of Processing Training
- Active tACS plus sham SoP (Active Comparator): Active alpha range tACS plus sham Speed of Processing Training
  Interventions: Device: alpha tACS
- Sham tACS plus active SoP (Active Comparator): Sham alpha range tACS plus Speed of Processing Training
  Interventions: Behavioral: Speed of Processing Training

INTERVENTIONS:
Device: alpha tACS — 2mA α-tACS (based on the IAF) over the prefrontal cortex (PFC)
  Arms: Active tACS plus active SoP; Active tACS plus sham SoP
Behavioral: Speed of Processing Training — SoP training will have a total of four conditions. In condition 1, participants will be asked to identity objects at increasingly brief exposures. For condition 2, identification of stimulus on the center of the screen will be requested from participants, while a second stimulus will appear somewhere in peripheral vision - stimulus duration, difficulty of the central localization task or the area in which targets may be located are used to change the level of difficulty. Condition 3 is similar to condition 2, but visual distractors are added. Finally, for condition 4, an auditory identification component is superimposed over the visual task (Jobe et al., 2001)
  Arms: Active tACS plus active SoP; Sham tACS plus active SoP

SUMMARY:
The current proposal aims to assess if the combination of Speed of Processing (SoP) training with alpha tACS (α-tACS) is able to increase brain speed of processing as assessed by the Useful Field of View (UFOV) when comparing to SoP training plus sham α-tACS. Moreover, a second aim is to assess if those changes in speed of processing transfer to other cognitive domains, such as memory, language and executive functioning. Furthermore, the mechanisms underlying these interventions will be tested, namely to assess brain connectivity and coherence as assessed by EEG. To that purpose, the aim of the current proposal is to conduct a double-blind, parallel randomized trial assessing the effects of combining SoP with alpha endogenous tACS (either active or sham) in participants with Mild Cognitive impairment (MCI).

DETAILED DESCRIPTION:
Dementia is thought to affect 6.3 million people across Europe and is especially prevalent in people over 85 years old (23.7%). In this sense, several cognitive training programs, alone or in combination with non-invasive brain stimulation have been used in order to ameliorate age-related cognitive impairments, and even to act in a prophylactic manner in order to prevent more extreme deficits, such as the ones presented in mild cognitive impairment, or even dementia.

Despite all these efforts, the effects of CT - combined or not - with several forms of non-invasive brain stimulation have been modest at most.

The current proposal aims to assess if Speed of Processing (SoP) training combined with alpha tACS (α-tACS) increases speed of processing as assessed by the Useful Field of View (UFOV) when comparing to SoP training and sham α-tACS. Furthermore, association betweens changes in speed of processing and changes in other cognitive domains, such as memory, language and executive functioning will be assessed. Finnaly, the current proposal aims at probing the mechanisms underlying these interventions, namely to test brain connectivity and coherence as assessed by EEG.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults aged 65 years and older, with cognitive complains in memory or other functions, which have declined over time

Exclusion Criteria:

* Score in the mini mental examination less than 23 (or over 28);
* Diagnosis of Alzheimer´s Disease, any other medical condition that may predispose participants for a forthcoming decline in function, or that may increase their risk of mortality during the duration of the study.
* Any contra-indication to tACS, severe sensory losses or communication difficulties that will prevent them from successfully complete the training.
* Had any cognitive training in the past.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Useful Field of View Test (UFOV) | Change from baseline to week 3
  UFOV is a measure of the speed of visual processing for rapid detection and localization of targets under conditions of divided visual attention and in the presence and absence of visual clutter at an above chance level (i.e. 75%).
Useful Field of View (UFOV) | Change from baseline to week 6
  UFOV is a measure of the speed of visual processing for rapid detection and localization of targets under conditions of divided visual attention and in the presence and absence of visual clutter at an above chance level (i.e. 75%).

SECONDARY OUTCOMES:
Executive Composite Score from the Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (NIH EXAMINER) | Change from baseline to week 3
  The NIH examiner executive composite comprises cognitive control, verbal fluency, and working memory assessments. Scores are based on the Item Response theory (IRT), which allows for the contribution of each item score is weighted by how effective that item measures that ability in any part of the continuum. Instead of a maximum or a minimum, higher scores, mean better performance.
Executive Composite Score from the Executive Abilities: Measures and Instruments for Neurobehavioral Evaluation and Research (NIH EXAMINER) | Change from baseline to week 6
  The NIH examiner executive composite comprises cognitive control, verbal fluency, and working memory assessments. Scores are based on the Item Response theory (IRT), which allows for the contribution of each item score is weighted by how effective that item measures that ability in any part of the continuum. Instead of a maximum or a minimum, higher scores, mean better performance.
EEG power in the alpha band | Change from baseline to week 3
  Total Power
EEG power in the alpha band | Change from baseline to week 6
  Total Power
P300 Event related potential - A | Change from baseline to week 3
  Amplitude of the P300 potential
P300 Event related potential - L | Change from baseline to week 3
  Latency of the P300 potential
P300 Event related potential - A | Change from baseline to week 6
  Amplitude of the P300 potential
P300 Event related potential - L | Change from baseline to week 6
  Latency of the P300 potential

OTHER OUTCOMES:
Useful Field of View (UFOV) | Change from baseline to 1 month follow-up (after intervention ended)
  Measure of the speed of visual processing for rapid detection and localization of targets under conditions of divided visual attention and in the presence and absence of visual clutter at an above chance level (i.e. 75%).
Useful Field of View (UFOV) | Change from baseline to 3 months follow-up (after intervention ended)
  Measure of the speed of visual processing for rapid detection and localization of targets under conditions of divided visual attention and in the presence and absence of visual clutter at an above chance level (i.e. 75%).
Useful Field of View (UFOV) | Change from baseline to 6 months follow-up (after intervention ended)
  Measure of the speed of visual processing for rapid detection and localization of targets under conditions of divided visual attention and in the presence and absence of visual clutter at an above chance level (i.e. 75%).
Executive Composite Score from NIH EXAMINER | Change from baseline to 1 month follow-up (after intervention ended)
  The NIH examiner comprises cognitive control, verbal fluency, and working memory assessments
Executive Composite Score from NIH EXAMINER | Change from baseline to 3 months follow-up (after intervention ended)
  The NIH examiner comprises cognitive control, verbal fluency, and working memory assessments
Executive Composite Score from NIH EXAMINER | Change from baseline to 6 months follow-up (after intervention ended)
  The NIH examiner comprises cognitive control, verbal fluency, and working memory assessments

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Leite, PhD, Principal Investigator — Portucalense University
Locations (1):
- Portucalense University, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Deidentified and coded data will be available to researchers upon request
Supporting Information: SAP
Time Frame: Data will be available upon study completion.
Access Criteria: Upon request.

REFERENCES:
- [Background] Jobe JB, Smith DM, Ball K, Tennstedt SL, Marsiske M, Willis SL, Rebok GW, Morris JN, Helmers KF, Leveck MD, Kleinman K. ACTIVE: a cognitive intervention trial to promote independence in older adults. Control Clin Trials. 2001 Aug;22(4):453-79. doi: 10.1016/s0197-2456(01)00139-8. PMID 11514044
- [Derived] Leite J, Goncalves OF, Carvalho S. Speed of Processing (SoP) Training Plus alpha-tACS in People With Mild Cognitive Impairment: A Double Blind, Parallel, Placebo Controlled Trial Study Protocol. Front Aging Neurosci. 2022 Jul 14;14:880510. doi: 10.3389/fnagi.2022.880510. eCollection 2022. PMID 35928993